CLINICAL TRIAL: NCT04777409
Title: A Randomised Double-blind Placebo-controlled Clinical Trial Investigating the Effect and Safety of Oral Semaglutide in Subjects With Early Alzheimer´s Disease (EVOKE Plus)
Brief Title: A Research Study Investigating Semaglutide in People With Early Alzheimer's Disease (EVOKE Plus)
Acronym: EVOKE Plus
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6535-4725; U1111-1259-2920 (Other: World Health Organization (WHO)); 2023-506918-45 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Early Alzheimer´s Disease
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral semaglutide (Experimental): Participants are given oral semaglutide once daily
  Interventions: Drug: Semaglutide
- Placebo (semaglutide) (Placebo Comparator): Participants are given oral placebo once daily
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Oral semaglutide once-daily, dose gradually increased to 14 mg. The study will last for up to 173 weeks
  Arms: Oral semaglutide
Drug: Placebo (semaglutide) — Oral placebo (semaglutide) once-daily. The study will last for up to 173 weeks
  Arms: Placebo (semaglutide)

SUMMARY:
This study is done to find out whether the medicine, semaglutide, has a positive effect on early Alzheimer's disease.

Participants will either get semaglutide or placebo (a "dummy" medicine which does not contain any study medicine) - which treatment participants get is decided by an equal chance.

The study will last for up to 173 weeks (about 3 years and 4 months). Participants will have 17 clinic visits and 1 phone call with the study doctor. The study includes various tests and scans. At 10 of the clinic visits participants will have blood samples taken.

Participants must have a study partner, who is willing to take part in the study.

Women cannot take part if pregnant, breastfeeding or plan to become pregnant during the study period.

A cerebrospinal fluid (CSF) sub-study will be performed as a part of the study. The sub-study will be performed on a selection of sites based on their experience with CSF sampling and willingness to participate in this sub-study. The endpoints related to this sub-study are exploratory only.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 55-85 years (both inclusive) at the time of signing informed consent.
* MCI (mild cognitive impairment) or mild dementia of the Alzheimer's type according to the NIA-AA (National Institute of Aging-Alzheimer's Association) 2018 criteria.
* CDR (Clinical Dementia Rating) global score of 0.5 and CDR of 0.5 or more in at least one of the three instrumental activities of daily living categories (personal care, home & hobbies, community affairs) Or CDR global score of 1.0
* RBANS (Repeatable Battery for the Assessment of Neuropsychological Status) delayed memory index score of below or equal to (≤) 85
* MMSE (Mini-Mental State Examination) greater than or equal to (≥) 22
* Amyloid positivity established with either amyloid PET (positron emission tomography), CSF (cerebrospinal fluid) Aβ1-42 or CSF Aβ1-42/Aβ1-40.
* If receiving an approved Alzheimer's disease treatment (such as acetylcholinesterase inhibitors, memantine or aducanumab) the dose must have been stable for at least 3 months prior to screening and should not be changed during the study unless medically necessary.

Exclusion Criteria:

* Brain Magnetic resonance imaging (MRI) (or Computed Tomography (CT)) scan suggestive of clinically significant structural CNS (central nervous system) disease confirmed by central read (e.g. cerebral large-vessel disease [large vessel (cortical) infarcts greater than (>) 10 milimeter (mm) in diameter], prior macro-haemorrhage [greater than 1 cubic centimetre (cm^3)], cerebral vascular malformations, cortical hemosiderosis, intracranial aneurism(s), intracranial tumours, changes suggestive of normal pressure hydrocephalus).
* Brain MRI (or CT) scan suggestive of strategic infarcts defined as bilateral thalamic lacunar infarcts and singular paramedian thalamic infarcts confirmed by central read.
* Evidence of a relevant neurological disorder other than mild cognitive impairment (MCI) or mild dementia of the Alzheimer's type at screening, including but not limited to Parkinson's disease, Lewy body disease, frontotemporal dementia of any type, Huntington's disease, amyotrophic lateral sclerosis, multiple sclerosis, systemic lupus erythematosus, progressive supranuclear palsy, neurosyphilis, human immunodeficiency virus (HIV), learning disability, intellectual disability, hypoxic cerebral damage, or significant head trauma with loss of consciousness that led to persistent cognitive deficits.
* Evidence of a clinically relevant or unstable psychiatric disorder, based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria, including schizophrenia or other psychotic disorder, or bipolar disorder. A participant with a history of major depression who has not had an episode in the last 24 months before the day of screening and is considered in remission or whose depression is controlled with treatment can be included in the study per investigator's judgement.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1840 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Change in the Clinical Dementia Rating - Sum of Boxes (CDR-SB) score | From baseline (week 0) to week 104
  Score on scale (0 to 18)
  Measures the impact of cognitive decline on daily function using the following six domains commonly affected in Alzheimer's disease:
  * Cognitive domains: memory, orientation, and judgement and problem solving
  * Function domains: community affairs, home and hobbies, and personal care Based on clinical information obtained from the subject and informant, an individual box score ranging from 0 to 3 is determined that represents "none" to "severe" impairment for each of the six domains.
  The CDR-Sum of Boxes (CDR-SB) score will be derived by adding the individual scores of the six domains at a given time point. The total CDR-SB score ranges from 0 to 18 with higher scores representing greater impairment.

SECONDARY OUTCOMES:
Main Phase: Change in the 24-item Alzheimer's Disease Cooperative Study Activities of Daily Living Scale for Mild Cognitive Impairment (ADCS-ADL-MCI) score | From baseline (week 0) to week 104
  Score on scale (0 to 53). An interview-based assessment of information provided by the study partner (informant). The total scores based on 18 items on the scale range from 0 to 53 with lower scores representing greater impairment.
Extension phase: Change in the ADCS-ADL-MCI score | From baseline (week 0) to week 156
  Score on scale (0 to 53) An interview-based assessment of information provided by the study partner (informant). The total scores based on 18 items on the scale range from 0 to 53 with lower scores representing greater impairment.
Main Phase: Time to progression to Clinical Dementia Rating (CDR) global score greater than or equal to (≥)1.0 among patients with CDR global score equal to (=) 0.5 at baseline | From baseline (week 0) up to week 156
  Week(s)
Extension Phase: Time to progression to Clinical Dementia Rating (CDR) global score greater than or equal to (≥)1.0 among patients with CDR global score equal to (=) 0.5 at baseline | From baseline (week 0) to week 156
  Week(s)
Main Phase: Change in the 13-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog-13) score | From baseline (week 0) to week 104
  Score on scale (0 to 85) Measures the severity of cognitive impairment in various domains including memory, language, orientation, praxis and executive function. The total scores on the scale range from 0 to 85 with higher scores representing greater impairment.
Extension Phase: Change in the 13-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog-13) score | From baseline (week 0) to week 156
  Score on scale (0 to 85) Measures the severity of cognitive impairment in various domains including memory, language, orientation, praxis and executive function. The total scores on the scale range from 0 to 85 with higher scores representing greater impairment.
Main Phase: Change in the Montreal Cognitive Assessment (MoCA) score | From baseline (week 0) to week 104
  Score on scale (0 to 30) The assessment includes 8 domains of cognitive function with total scores ranging from 0 to 30 and lower scores indicating greater impairment.
Extension Phase: Change in the Montreal Cognitive Assessment (MoCA) score | From baseline (week 0) to week 156
  Score on scale (0 to 30) The assessment includes 8 domains of cognitive function with total scores ranging from 0 to 30 and lower scores indicating greater impairment.
Main Phase: Change in the Alzheimer's Disease Composite Score (ADCOMS) | From baseline (week 0) to week 104
  Score on scale (0 to 1.97) The ADCOMS is a composite clinical outcome comprising 4 items from the ADAS-Cog-13, 2 items from the MMSE and all 6 items from the CDR-SB.32 The total scores on the scale range from 0 to 1.97 with higher scores indicating greater impairment.
Extension Phase: Change in the Alzheimer's Disease Composite Score (ADCOMS) | From baseline (week 0) to week 156
  Score on scale (0 to 1.97) The ADCOMS is a composite clinical outcome comprising 4 items from the ADAS-Cog-13, 2 items from the MMSE and all 6 items from the CDR-SB.32 The total scores on the scale range from 0 to 1.97 with higher scores indicating greater impairment.
Main Phase: Change in the Mini-Mental State Examination (MMSE) score | From baseline (week 0) to week 104
  Score on scale (0 to 30) The MMSE measures orientation, attention, memory, language and visuo-spatial function. The total scores on the scale range from 0 to 30 with lower scores indicating greater impairment.
Extension Phase: Change in the Mini-Mental State Examination (MMSE) score | From baseline (week 0) to week 156
  Score on scale (0 to 30) The MMSE measures orientation, attention, memory, language and visuo-spatial function. The total scores on the scale range from 0 to 30 with lower scores indicating greater impairment.
Main Phase: Time to progression in disease stage based on CDR global score | From baseline (week 0) up to week 156
  Week(s)
Extension Phase: Time to progression in disease stage based on CDR global score | From baseline (week 0) to week 156
  Week(s)
Main Phase: Change in the composite Z-score based on the three outcome measures CDR-SB, ADCS-ADL-MCI, and ADAS-Cog-13 | From baseline (week 0) to week 104
  Score
Extension Phase: Change in the composite Z-score based on the three outcome measures CDR-SB, ADCS-ADL-MCI, and ADAS-Cog-13 | From baseline (week 0) to week 156
  Score
Main Phase: Change in the 10-item Neuropsychiatric Inventory (NPI) score | From baseline (week 0) to week 104
  104 Score on scale (0 to 120) The 10-item scale assesses symptoms including delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability and aberrant motor activity. For each domain the frequency (4-point scale) and severity (3-point scale) of symptoms is reported. The score for each domain is calculated by multiplying the frequency and severity score. The total 10-item NPI score is 0 to 120 with higher scores indicating a greater symptomatology.
Extension Phase: Change in the 10-item Neuropsychiatric Inventory (NPI) score | From baseline (week 0) to week 156
  104 Score on scale (0 to 120) The 10-item scale assesses symptoms including delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability and aberrant motor activity. For each domain the frequency (4-point scale) and severity (3-point scale) of symptoms is reported. The score for each domain is calculated by multiplying the frequency and severity score. The total 10-item NPI score is 0 to 120 with higher scores indicating a greater symptomatology.
Main Phase: Change in high sensitivity C-reactive protein level | From baseline (week 0) to week 104
  Ratio to baseline
Extension Phase: Change in high sensitivity C-reactive protein level | From baseline (week 0) to week 156
  Ratio to baseline
Main Phase: Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) up to week 156
  Number of events
Extension Phase: Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to week 156
  Number of events
Main Phase: Time to first occurrence of major adverse cardiovascular event (MACE) comprising non-fatal myocardial infarction, non-fatal stroke and allcause death | From baseline (week 0) to week 104
  Week(s)
Extension Phase: Time to first occurrence of major adverse cardiovascular event (MACE) comprising non-fatal myocardial infarction, non-fatal stroke and allcause death | From baseline (week 0) to week 156
  Week(s)
Main Phase: Time to first occurrence of stroke | From baseline (week 0) to week 104
  Weeks
Extension Phase: Time to first occurrence of stroke | From baseline (week 0) to week 156
  Weeks
Main Phase: Change in the EQ-5D-5L (proxy version) index score | From baseline (week 0) to week 104
  Score The EQ-5D-5L descriptive system comprises mobility, self-care, usual activities, pain/discomfort and anxiety/depression with five response levels each (no problems, slight problems, moderate problems, severe problems, unable to /extreme problems). The EQ-5D-5L proxy version 1 (the study partner is asked to rate how he/she [the proxy] would rate the subject´s health) will be used in this trial.
Extension Phase: Change in the EQ-5D-5L (proxy version) index score | From baseline (week 0) to week 156
  Score The EQ-5D-5L descriptive system comprises mobility, self-care, usual activities, pain/discomfort and anxiety/depression with five response levels each (no problems, slight problems, moderate problems, severe problems, unable to /extreme problems). The EQ-5D-5L proxy version 1 (the study partner is asked to rate how he/she [the proxy] would rate the subject´s health) will be used in this trial.
Extension phase: Change in the CDR-SB score | From baseline (week 0) to week 156
  Score on scale (0 to 18)
  Measures the impact of cognitive decline on daily function using the following six domains commonly affected in Alzheimer's disease:
  * Cognitive domains: memory, orientation, and judgement and problem solving
  * Function domains: community affairs, home and hobbies, and personal care Based on clinical information obtained from the subject and informant, an individual box score ranging from 0 to 3 is determined that represents "none" to "severe" impairment for each of the six domains.
  The CDR-Sum of Boxes (CDR-SB) score will be derived by adding the individual scores of the six domains at a given time point. The total CDR-SB score ranges from 0 to 18 with higher scores representing greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (486):
- United States (107):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Imaging Endpoints, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Tucson Neuroscience Research, Tucson, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - ASCLEPES Research Centers,, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA_Los Angeles, Los Angeles, California
  - Wr-Pri, Llc, Newport Beach, California
  - Well Care Medical Center, Panorama City, California
  - Cedars-Sinai Medical Center, Pasadena, California
  - Sharp Neurocog Res Ctr, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Calfornia Neurosc Resrch Med, Sherman Oaks, California
  - Southern California Research LLC, Simi Valley, California
  - Mountain Neurological Research Center, Inc., Basalt, Colorado
  - Denver Neurological Research, Denver, Colorado
  - Mile High Research Center, Denver, Colorado
  - Nuvance Health, Associtd Neuro, Danbury, Connecticut
  - Yale University, Fairfield, Connecticut
  - Research Center for Clinical Studies, Inc, Norwalk, Connecticut
  - Topaz Clinical Research, Apopka, Florida
  - JEM Research Institute, Atlantis, Florida
  - Visionary Investigators Network, Aventura, Florida
  - K2 Medical Research - Winter Garden, Clermont, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Integrity Clinical Research, LLC, Doral, Florida
  - Neuropsychiatric Research Cent, Fort Myers, Florida
  - Finlay Medical Research Group, Greenacres City, Florida
  - Indago Research & Health Center Inc., Hialeah, Florida
  - Hlth Cr Family Rehab & Res Ctr, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - K2 The Villages, Lady Lake, Florida
  - K2 Medical Research, Maitland, Maitland, Florida
  - Hlth Cr Family Rehab & Res Ctr, Miami, Florida
  - Premier Clin Res Inst, Inc., Miami, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Central Miami Medical Institute, Miami, Florida
  - Novel Clinical Research Center, LLC, Miami, Florida
  - IMIC, Inc- Medical Research, Miami, Florida
  - The Neurology Research Group, Miami, Florida
  - Visionary Inv Ntwrk_Miami, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Suncoast Clin Res Port Richey, New Port Richey, Florida
  - Suncoast Clinical Research, Inc._New Port Richey, New Port Richey, Florida
  - K2 Medical Research - Winter Garden, Ocoee, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - The Roskamp Institute, Inc., Sarasota, Florida
  - Brain Matters Resrch Kane Cntr, Stuart, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Stedman Clinical Trials LLC, Tampa, Florida
  - Palm Beach Neuro Premiere Res, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Hawaii Neuroscience, Memory Disorders Center, Honolulu, Hawaii
  - Velocity Clinical Research, Meridian, Meridian, Idaho
  - Velocity Clinical Research, Meridian, Idaho
  - Josephson Wallack Munshower, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - University of Kentucky_Lexington_0, Lexington, Kentucky
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - ActivMed Practice & Research LLC, Methuen, Massachusetts
  - Bronson Lakeview Neurobehavioral Health, Paw Paw, Michigan
  - HealthPartners Center for Memory and Aging, Saint Paul, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Altea Research Institute, Las Vegas, Nevada
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Patient First MD,clinical Trials, Middletown, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Albuquerque neuroscience Inc, Albuquerque, New Mexico
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurological Assoc Long Island, Lake Success, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - NYU Grossman School of Med, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - SUNY Upstate Medical University_Syracuse, Syracuse, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - AMC Research, LLC, Matthews, North Carolina
  - NeuroScience Research Center, LLC, Canton, Ohio
  - Valley Medical Primary Care, Centerville, Ohio
  - Insight Clinical Trials LLC, Independence, Ohio
  - Cleveland Clinic_Lakewood, Lakewood, Ohio
  - Central States Research, LLC, Tulsa, Oklahoma
  - Summit Research Network Oregon Inc., Portland, Oregon
  - Neural Net Research, LLC, Portland, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Lowcountry Center for Vet Res, Charleston, South Carolina
  - Coastal Neurology, Port Royal, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Genesis Neuroscience Clinic, Knoxville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Neurology Consultants of Dallas, Dallas, Texas
  - Balyor College of Medicine, Houston, Texas
  - Univ Of Texas Hlth Science Cntr, Houston, Texas
  - Mt. Olympus Medical Research, Katy, Texas
  - Glenn Biggs Inst-Alzhm Neuro, San Antonio, Texas
  - Shirzadi Shahin, MD, Sugar Land, Texas
  - Memory Clinic, Inc, Bennington, Vermont
  - Integrated Neurology Services, Falls Church, Virginia
  - Booth Gardner Parkinson's Cre, Kirkland, Washington
  - Harborview Medical Center, Seattle, Washington
- Argentina (7):
  - Instituto Medico Especializado_Capital Federal, Ciudad de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Metabolicas (IDIM), Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Clínica Nuestra Señora de las Nieves, CABA
  - FLENI, CABA
  - Instituto Privado Kremer, Córdoba
  - Fundación Scherbovsky, Mendoza
- Australia (10):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - HammondCare Greenwich, Greenwich, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - KaRa Institute of Neurological Disease Pty Ltd, Macquarie Park, New South Wales
  - Hunter New England Local Health District - Neuropsychiatry, Waratah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Medical and Cognitive Research Unit - Austin Health, Ivanhoe, Victoria
  - HammondCare, Malvern, Victoria
  - Alzheimer's Research Australia, Nedlands, Western Australia
  - Australian Alzheimer's Research Foundation Incorporated, Nedlands, Western Australia
- Austria (5):
  - Universitätsklinik für Neurologie, Graz
  - LKH-Univ. Kliniken Innsbruck, Innsbruck
  - Medizinische Univ. Innsbruck, Innsbruck
  - Univ. Klinik für Neurologie, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (6):
  - AZ Sint-Jan - Campus Sint-Jan - Neurology, Bruges
  - UZA - UZ Antwerpen - Department of Neurology, Edegem
  - UZ Gent - Neurologie, Ghent
  - AZ Groeninge - Kortrijk - Neurologie, Kortrijk
  - UZ Leuven - Geheugenkliniek, Leuven
  - Clinique CHC MontLégia - Service Neurologie, Liège
- Brazil (10):
  - L2 IP Instituto de Pesquisas Clinicas Ltda, Brasília, Federal District
  - Hospital das Clínicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Clinica Clinilive Ltda, Maringá, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - BR Trials - Ensaios Clínicos e Consultoria Ltda., São Paulo, São Paulo
  - Assoc. Paulista para o Desenvolvimento da Medicina - UNIFESP, São Paulo, São Paulo
  - Sociedade Beneficente Israelita Bras Hosp Albert Einstein, São Paulo, São Paulo
  - Centro de Psiquiatria Sandra Rushel, Rio de Janeiro
- Bulgaria (5):
  - "MHATNP "Sv. Naum"" EAD, Sofia
  - MHATNP Sveti Naum EAD, Sofia
  - DCC Sv. Vrach and Sv. Sv. Kuzma and Damyan OOD, Psychiatry, Sofia
  - "UMHAT "Aleksandrovska", Neurology clinic, Sofia
  - MMA, MHAT-Sofia, Neurology clinic, Sofia
- Canada (18):
  - OCT Research ULC (dba Okanagan Clinical Trials), Kelowna, British Columbia
  - Medical Arts Health Research Group, North Vancouver, British Columbia
  - Medical Arts Health Research Group_Kelowna, Penticton, British Columbia
  - Island Health (Research and Capacity Building), Victoria, British Columbia
  - True North Clinical Research - Halifax, Halifax, Nova Scotia
  - True North Clinical Research - New Minas, New Minas, Nova Scotia
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Recherches Neuro-Hippocampe Inc, Ottowa, Ontario
  - Kawartha Centre Redefining Healthy Aging, Peterborough, Ontario
  - Memory Program, Toronto, Ontario
  - Centricity Research LMC, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - MoCA Research Innovation Inc, Greenfield Park, Quebec
  - Douglas Hosp Res Ctr, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- China (36):
  - Beijing Chao-Yang Hospital, Capital Medical University-Neuro, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University-Neurology, Beijing, Beijing Municipality
  - Beijing Hospital-Neurology, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University-Neurology, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University-Neurology Center, Beijing, Beijing Municipality
  - Beijing Anding Hospital Capital Medical University-Geriatric Psychiatry, Beijing, Beijing Municipality
  - Peking University Sixth Hospital-Geriatrics, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital-Geriatrics, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital-Neurology, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University-Geriatrics, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital-Neurology, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University-Neurology, Guangzhou, Guangdong
  - Guangzhou First People's Hospital-Neurology, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University-Neurology, Guangzhou, Guangdong
  - The Affiliated Brain Hospital of Guangzhou Medical University-Neurology, Guangzhou, Guangdong
  - Henan Provincial People's Hospital-Neurology, Zhengzhou, Henan
  - Xiangya Hospital Central South University-Neurology, Changsha, Hunan
  - Baogang Hospital of Inner Mongolia-Neurology, Baotou, Inner Mongolia
  - Nanjing Brain Hospital-Neurology, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital-Neurology, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University-Nephrology, Nanjing, Jiangsu
  - Wuxi Mental Health Center-Psychiatry, Wuxi, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Northern Jiangsu People's Hospital-Neurology, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University-Neurol, Nanchang, Jiangxi
  - The first Bethune Hospital of Jilin University, Neurology, Changchun, Jilin
  - The First Bethune Hospital of Jilin University-Neurology, Changchun, Jilin
  - Qinghai Provincial People's Hospital-Geriatrics, Xining, Qinghai
  - Huashan Hospital Fudan University-Neurology, Shanghai, Shanghai Municipality
  - Dongfang Hospital Affiliated to Shanghai Tongji University-Neurology, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hosp. Affili. to SHJT Univer-Neurology, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University-Neurology, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University-Mental health center, Chengdu, Sichuan
  - General Hospital of Tianjin Medical University-Neurology, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital-Neurology, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine-Neurology, Hangzhou, Zhejiang
- Croatia (4):
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - KBC Zagreb, Klinika za neurologiju, Zagreb
  - KBC Zagreb_Neurology, Zagreb
  - Poliklinika Bonifarm, Zagreb
- Czechia (6):
  - Neuro Health Centrum s.r.o., Brno-Líšeň
  - NeuroHK s.r.o., Choceň
  - AGE Centrum, Olomouc
  - AD71 s.r.o., Prague
  - Neuropsychiatrie s.r.o., Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- Denmark (3):
  - Aarhus Universitetshospital - Neurologisk Klinik, Aarhus N
  - Rigshospitalet - afsnit 8015 Hukommelsesklinikken, København Ø
  - Sjællands Universitetshospital_Roskilde, Roskilde
- Finland (3):
  - CRST Helsinki, Helsinki
  - Aivotutkimusyksikkö, Kuopio
  - CRST Turku, Turku
- France (14):
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Pellegrin, Bordeaux
  - Hospices Civils de Lyon-Hopital Pierre Wertheimer, Bron
  - Centre Hospitalier Universitaire de Dijon-Hopital Le Bocage, Dijon
  - Centre Hospitalier Universitaire de Lille-Hopital Roger Salengro, Lille
  - Centre Hospitalier Et Universitaire de Limoges-Hopital Dupuytren, Limoges
  - Assistance Publique Hopitaux de Marseille-Hopital de La Timone-1, Marseille
  - Centre Hospitalier Universitaire de Nice-Institut Claude Pompidou, Nice
  - Aphp-Hopital Lariboisiere-1, Paris
  - Aphp-Hopital La Pitie Salpetriere-3, Paris
  - Chu de Reims-Hopital Maison Blanche, Reims
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-2, Saint-Herblain
  - Les Hopitaux Universitaires de Strasbourg-Hopital de La Robertsau, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse-Hopital La Grave, Toulouse
  - Hospices Civils de Lyon-Hopital Des Charpennes, Villeurbanne
- Germany (2):
  - Universitätsklinikum Köln - Klinik und Poliklinik für Psychiatrie und Psychotherapie, Cologne
  - Universitätsklinikum Münster - Neurologie, Münster
- Greece (8):
  - Naval Hospital of Athens, Athens
  - Henry Dunant Hospital Center,2nd Neurological Department, Athens
  - Aiginitio Hospital, 1st Neurology Clinic, Athens
  - "Hygeia" General Hospital of Athens, Memory clinic, Athens
  - University General Hospital of Athens "Attiko", Chaidari, Athens
  - Iatriko Athinon (Athens Medical Center),Memory Disorders Cli, Marousi
  - AHEPA General University Hospital, Thessaloniki
  - EUROMEDICA General Clinic of Thessaloniki,Neurology Dpt, Thessaloniki
- Hungary (12):
  - Clinexpert Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Semmelweis Egyetem ÁOK, Budapest
  - DE Kenézy Gyula Campus, Pszichiátriai és Pszichoterápiai Klinika, Debrecen
  - DE Gyógyszerfejlesztési Koordinációs Központ Pszichiátria, Debrecen
  - Bugát Pál Kórház, Gyöngyös
  - Petz Aladar Megyei Korhaz, Győr
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - DR. MÁTHÉ ÉS TÁRSA Egészségügyi és Szolgáltató Betéti Társaság, Kalocsa
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Psychotech Kft., Pécs
  - Szent Borbála Kórház, Tatabánya
  - Belvárosi Egészségház Kft., Zalaegerszeg
- Ireland (5):
  - Mercy Hospital Cork, Cork
  - St Vincent's Neurology Dept, Dublin
  - St Vincent's University Hospital, Dublin
  - Mercer's Institute for Successful Aging, Dublin
  - Tallaght University Hospital, Dublin
- Israel (4):
  - Rambam MC - The Stroke and Cognition Institute, Haifa
  - Rabin MC Beilinson - Cognitive Neurology Clinic, Petah Tikva
  - Sourasky MC - Cognitive Neurology Department, Tel Aviv
  - Sheba MC - Memory Clinic, Tel Hashomer, Ramat Gan
- Italy (14):
  - AOU Ospedali Riuniti S.O.D, Ancona
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Università degli studi G. D'Annunzio di Chieti - CAST - Neurologia, Chieti
  - AOU Careggi Firenze, Florence
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele Milano, Milan
  - ASST Monza e Brianza Ospedale San Gerardo, Monza
  - Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Pol. Uni. Campus Biomedico UOC Neurologia, Roma
  - Policlinico Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Neuroscienze, Organi di Senso e Torace, Roma
  - Fondazione Santa Lucia IRCCS, Roma
  - AOU Città della Salute e della Scienza di Torino, Torino
- Japan (59):
  - Iwaki Clinic_Psychosomatic medicine, Anan, Tokushima
  - Yachiyo Hospital_Neurology, Anjo-shi, Aichi
  - Abe Clinic, Arakawa-ku,Tokyo
  - Memory Clinic Ochanomizu, Bunkyo-ku, Tokyo
  - Institute of Science Tokyo Hospital_ Neurology, Bunkyo-ku,Tokyo
  - Tokyo Medical And Dental University Hospital, Bunkyo-ku,Tokyo
  - Kashiwado Hospital_Neurology, Chib-shi, Chiba
  - Kashiwado Hospital, Chib-shi, Chiba
  - Enomoto Internal Medicine Clinic, Chofu-shi,Tokyo
  - Shinozuka Hospital_Neurology, Fujioka-Shi, Gunma
  - P-one Clinic, Hachioji-shi, Tokyo
  - National Hospital Organization Tenryu Hospital, Hamamatsu-shi, Shizuoka
  - Hyogo Prefectural HarimaHimeji General Medical Center_Dept. of Aging Brain&Cognitive, Himeji-shi, Hyogo
  - Tsukazaki Hospital_Department of Neurology, Himeji-shi, Hyogo
  - Himeji Central Hospital Clinic, Himeji-shi, Hyogo
  - Hatsuta Neurology Clinic, Hirakata-Shi,Osaka
  - Imon Yukari Neurology Clinic, Hiroshima-shi, Hiroshima
  - Hikaru-kai Medical Corporation Hiroshima Neurology Clinic, Hiroshima-shi, Hiroshima
  - Hiroshima Neurology Clinic, Hiroshima-shi, Hiroshima
  - Nagamitsu Clinic, Hofu-shi, Yamaguchi
  - Ina Central Hospital_Neurology, Ina-shi, Nagano
  - Ina Central Hospital, Ina-shi, Nagano
  - Kawasaki Saiwai Clinic_Internal Medicine, Kanagawa
  - Kishiro Mental Clinic, Kawasaki-shi , Kanagawa
  - Koukan Clinic, Kawasaki-shi, Kanagawa
  - Teikyo Univ. HP, Mizonokuchi_Neurosurgery, Kawasaki-shi, Kanagawa
  - Teikyo University Hospital, Mizonokuchi_Kawasaki-shi, Kanagawa, Kawasaki-shi, Kanagawa
  - Kobe University Hospital_Neurology, Kobe-shi, Hyogo
  - Kobe University Hospital_Radiology, Kobe-shi, Hyogo
  - National Center of Neurology and Psychiatry_Neurology, Kodaira-shi, Tokyo
  - Southern Tohoku Medical Clinic, Koriyama-shi, Fukushima
  - Katayama Medical Clinic, Kurashiki-shi, Okayama
  - Nozomi Memory Clinic, Mitaka-shi,Tokyo
  - Kikukawa clinic, Nerima-ku, Tokyo
  - General Rehabilitation Center Midori Hospital_Neurology, Niigata-shi, Niigata
  - General Rehabilitation Center · Midori Hospital, Niigata-shi, Niigata
  - National Center for Geriatrics and Gerontology_Comprehensive care, Obu-shi, Aichi
  - OKAYAMA KYOKUTO HOSPITAL_Radiology, Okayama-shi, Okayama
  - Jichiidai Station Brain Clinic, Shimotsuke-shi, Tochigi
  - ALZCLINIC PET LAB_Radiology, Shinjuku-ku, Tokyo
  - Keio University Hospital_Neurology, Shinjuku-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Shizuoka City Shimizu Hospital_Neurology, Shizuoka-shi, Shizuoka
  - Kagawa Prefectural Central Hospital_Neurology, Takamatsu-shi, Kagawa
  - Kagawa Prefectural Central Hospital_Takamatsu-shi, Kagawa, Takamatsu-shi, Kagawa
  - Takatsuki General Hospital_Neurology, Takatsuki-Shi, Osaka
  - Saino Clinic, Tokorozawa-shi,Saitama
  - Itsuki Hospital_Neurology, Tokushima-shi, Tokushima
  - Alzclinic Tokyo, Tokyo
  - Tokyo Center Clinic, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center_psychiatry, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Kurumi CLINIC, Tokyo
  - ALZCLINIC PET LAB_Psychiatry, Tokyo
  - Tokyo Medical Univ. Hospital, Tokyo
  - Memory Clinic Toride, Toride-shi, Ibaraki
  - MI Clinic, Toyonaka-shi, Osaka
  - Medical Corporation Midorikai Wako Hospital_Psychiatry, Wako-shi, Saitama
  - Yuaikai Yuai Clinic, Yokohama-shi, Kanagawa
- Netherlands (4):
  - Brain Research Center, 's-Hertogenbosch
  - Amphia Ziekenhuis, Breda
  - Spaarne Gasthuis, Haarlem
  - Radboudumc, Nijmegen
- Poland (13):
  - Linden sp. z o.o. sp. k., Krakow, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska prof. Konrad Rejdak, Lublin, Lublin Voivodeship
  - Centrum Medyczne Neuromed, Bydgoszcz
  - Centrum Zdrowia Psychicznego Biomed, Kielce
  - Szpital Uniwersytecki w Krakowie od. Neurologii, Krakow
  - Centrum Neurologii Klinicznej, Krakow
  - Nzoz Neuromed, Lublin
  - INSTYTUT ZDROWIA DR BOCZARSKA-JEDYNAKSp. z o.o. Sp. k., Oświęcim
  - NZOZ NEURO - KARD Ilkowski i Partnerzy Sp. Part. Lekarzy, Poznan
  - Centrum Medyczne SENIOR, Sopot
  - Osrodek Alzheimerowski Sp. z o.o., Ścinawa
  - Centrum Medyczne Neuro Protect, Warsaw
  - NZOZ Wrocławskie Centrum Alzheimerowskie, Wroclaw
- Portugal (8):
  - ULS De Matosinhos E.P.E.- Hospital Pedro Hispano, Senhora Da Hora, Matosinhos, Matosinhos
  - ULS De Braga, E.P.E. - Hospital de Braga, Braga
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - ULS Do Alto Ave, E.P.E. - Hospital Senhora da Oliveira - Guimarães, Guimarães
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital Egas Moniz, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Campus Neurologico Senior (CNS) Saude Lda, Torres Vedras
- Romania (10):
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş, Mureș County
  - CMI Neurologie Dr Popa Izabela, Timișoara, Timiș County
  - Sana Monitoring SRL, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Cai Ferate Constanta, Constanța
  - Spitalul Clinic Judetean De Urgenta Sfantul Apostol Andrei Constanta, Constanța
  - Med Anima Iasi, Iași
  - CMI Dr. Buhaș Ramocea Elena Daniela - Cabinet Medical de Psihiarie, Oradea
  - Aria Clinic SRL, Sibiu
  - Centrul Medical Neuro Therapy, Timișoara
- Russia (18):
  - SAI of Health "Interregional Clinic Diagnostic Center", Kazan'
  - SAHI Kuzbass Hospital(former Regional clinical hospital), Kemerovo
  - Federal Siberian Research Clinical Center under FMBA of Rus, Krasnoyarsk
  - FSBI "Mental Health Research Center", Moscow
  - FSAEI 1st Moscow Federal Med University na Sechenov, Moscow
  - RMAPE, Moscow
  - Pirogov Russian National Research Medical University MoH, Moscow
  - Ezramed Clinic Llc, Omsk
  - Research Center for Treatment and Rehabilitation "Phoenix", Rostov-on-Don
  - Psychiatric hospital of st. Nicholas the wonderworker, Saint Petersburg
  - N.-E. State Medical University n.a. Mechnikov, Saint Petersburg
  - S.M. Kirov Military Medical Academy,Depart.&Clinic Nerv Dis, Saint Petersburg
  - SHI "Saratov City Clinical Hospital #2 n.a. V.Razumovskij", Saratov
  - Center of Clinica Trials "Nebbiolo", Tomsk
  - LLC "Clinic Stolet", Tomsk
  - National medical holdiNational medical holding "Medstandard", Ufa
  - SAHI SR "Sverdlovsk Regional Clinical Psychiatric Hospital", Yekaterinburg
  - Joint Stock Company "Medical technologies", Yekaterinburg
- Serbia (3):
  - Neurology clinic, University Clinical Center of Serbia, Belgrade
  - Special Hospital for Psychiatric Disorders "Kovin", Kovin
  - University clinical center of Vojvodina, Neurology clinic, Novi Sad
- Slovakia (5):
  - I. neurologicka klinika LF UK a UNB, Bratislava
  - Psychiatricka klinika LF UK a UNB, Bratislava
  - Neurologicka klinika UPJS LF a UNLP, Košice
  - NEURES, neurologicka ambulancia, Krompachy
  - Crystal Comfort s.r.o., Vranov nad Topľou
- Slovenia (3):
  - UKC Ljubljana, Department of Neurology, Ljubljana
  - UKC Maribor - neurology, Maribor
  - Private Neurology Practice - Nova Gorica, Nova Gorica
- South Africa (7):
  - Excellentis Clinical Trial Consultants, George, Eastern Cape
  - IATROS International, Bloemfontein, Free State
  - Dr Stanley Lipschitz Clinic Inc, Johannesburg, Gauteng
  - Denmar Psychiatric Hospital, Pretoria, Gauteng
  - ACF Neurological service, Cape Town, Western Cape
  - Flexivest Fourteen Research Centre, Cape Town, Western Cape
  - Cape Trial Centre, Cape Town, Western Cape
- South Korea (14):
  - MyongJi Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Hanyang University Medical Center, Seoul
  - Hanyang university seoul hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center_Seoul, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundación ACE, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Doctor Peset, Valencia
- Sweden (3):
  - Minnesmottagning specialiserad Malmö, Malmo
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - Geriatriskt centrum, Umeå, Umeå
- Switzerland (4):
  - Spitalzentrum Biel, Biel/Bienne
  - Centre de la Mémoire, Geneva
  - Centre Leenaards de la mémoire CHUV, Lausanne
  - Klinik für Neurologie Kantonsspital St.Gallen, Sankt Gallen
- Taiwan (10):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaoshiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital_main, Taipei
  - Taipei Veteran General Hospital_Dept of Neurology, Taipei
  - Taipei Veteran General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Turkey (Türkiye) (12):
  - Hacettepe University Medical Faculty Hospital, Altindag/Ankara
  - Hacettepe Üniversitesi Hastanesi- Nöroloji, Altindag/Ankara
  - Dokuz Eylül Üniversitesi Araştırma Uygulama Hastanesi- Nöroloji, Balcova / Izmir
  - Eskisehir Osmangazi University Sağlık Uygulama ve Arastirma, Eskişehir
  - Eskişehir Osmangazi Üniversitesi Hastanesi- Nöroloji, Eskişehir
  - Istanbul Bezmi Alem Vakif University Tip Faculty Hospital, Istanbul
  - Istanbul University Medical Faculty Neurology Department, Istanbul
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Hastanesi- Nöroloji, Istanbul
  - Izmir Economics University Medical Point Hospital Neurology D, Izmir
  - İzmir Ekonomi Üniversitesi Medicalpoint Hastanesi-Nöroloji, Izmir
  - Ondokuz Mayis University Saglik Uygulama ve Arastirma Merkez, Samsun
  - Ondokuz Mayıs Üniversitesi Hastanesi- Nöroloji, Samsun
- Ukraine (10):
  - Chernivtsi Emergency Hospital - Center of Emergency Neurology, Chernivtsi
  - Medical Center 'Neiron', Kharkiv
  - Medical Centre 'Neiron', Kharkiv
  - Chebotarev Institute of Gerontology of NAMSU - Age Physiology and Pathology department, Kyiv
  - Volyn Regional Clinical Hospital - Neurology department, Lutsk
  - Main Unit of 'Odesa Regional Medical Centre for Mental Health' - Department 18, Odesa
  - Odesa Regional Medical Center for Mental Health, Odesa
  - Sumy Regional Clinical Hospital - Neurology department, Sumy
  - Medical Centre 'SALUTEM' - Medical and preventive care department, Vinnytsia
  - Zaporizhia Regional Clinical Hospital - Department of neurology No. 1, Zaporizhzhia
- United Kingdom (16):
  - Fritchie Centre, Cheltenham, Gloucestershire
  - Royal Cornhill Hospital, Aberdeen
  - RICE - The Research Institute for the Care of Older People, Bath
  - Dementia Research Unit,, Crowborough
  - Dementia Research Unit, Crowborough
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - St Pancras Clinical Research, London
  - St Georges Hospital, London
  - Imperial College London - Imperial College Memory Research Centre, London
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester
  - NeuroClin, Motherwell
  - Newcastle University, Newcastle upon Tyne
  - Warneford Hospital, Oxford
  - Moorgreen Hospital, Southampton
  - Kings Hill Research Centre, Swindon

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Scheltens P, Atri A, Feldman HH, Zetterberg H, Sano M, Johannsen P, Colombo TL, Bardtrum L, Jeppesen R, Hansen CT, Cummings JL. Baseline characteristics from evoke and evoke+: Two phase 3 randomized placebo-controlled trials of semaglutide in participants with early-stage symptomatic Alzheimer's disease. Alzheimers Dement (N Y). 2026 Jan 10;12(1):e70200. doi: 10.1002/trc2.70200. eCollection 2026 Jan-Mar. PMID 41522368
- [Derived] Cummings JL, Atri A, Feldman HH, Hansson O, Sano M, Knop FK, Johannsen P, Leon T, Scheltens P. evoke and evoke+: design of two large-scale, double-blind, placebo-controlled, phase 3 studies evaluating efficacy, safety, and tolerability of semaglutide in early-stage symptomatic Alzheimer's disease. Alzheimers Res Ther. 2025 Jan 8;17(1):14. doi: 10.1186/s13195-024-01666-7. PMID 39780249
- [Derived] van Sloten TT, Luchsinger JA, Launer LJ, Strachan M, Cukierman-Yaffe T, Gerstein HC, Sattar N, Biessels GJ. Call for effective therapies for preventing dementia in people with type 2 diabetes. Lancet Diabetes Endocrinol. 2024 Aug;12(8):510-513. doi: 10.1016/S2213-8587(24)00158-X. Epub 2024 Jun 17. No abstract available. PMID 38901446